CLINICAL TRIAL: NCT05026749
Title: Azithromycin Treatment for Respiratory Syncytial Virus-induced Respiratory Failure in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michele Kong, MD, PI, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300007862; 1R01HD105678-01 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; AZM; ICU; Respiratory Support; Children
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator)
  Interventions: Other: Control Group
- AZM 20mg/kg Treatment Group (Active Comparator)
  Interventions: Drug: AZM Group

INTERVENTIONS:
Drug: AZM Group — AZM at 20 mg/kg will be given intravenous daily for 3 days once patients are consented and enrolled into the study.
  Arms: AZM 20mg/kg Treatment Group
Other: Control Group — Saline will be given intravenous daily for 3 days once patients are consented and enrolled into the study.
  Arms: Control Group

SUMMARY:
The overarching hypothesis of the ARRC trial is that administration of Azithromycin (AZM) during acute, Respiratory Syncytial Virus (RSV)-induced respiratory failure will be beneficial, mediated through the matrix metalloproteinase (MMP)-9 pathway.

DETAILED DESCRIPTION:
The proposed study will be a randomized, double-blinded, placebo-controlled Phase III trial to examine the efficacy of AZM therapy relative to placebo in reducing RSV-related morbidity. Patients will be recruited during acute hospitalization and admission to the ICU at 10 pediatric hospitals. The target population selected is pediatric patients with severe RSV lung disease as defined by need for ICU management and intensive respiratory support.

ELIGIBILITY:
Inclusion criteria:

* Admission to the pediatric ICU with a confirmed diagnosis of RSV infection. RSV infection is based on a positive nasal swab for RSV fluorescent antibody or via multiplex assay or culture;
* Requiring intensive respiratory support defined as either mechanical ventilation or NIV (BiPAP or CPAP) or HFNC (at >1 L/kg/min of flow
* Enrollment into the study within 48 hours of ICU admission and placement on intensive respiratory support;
* Onset of RSV-related symptoms must be less than 5 days
* Age: Neonates-2 years. For those less than 1 week of age, they must have been discharged home from the hospital after their birth.

Exclusion criteria:

* AZM use within 7 days of ICU admission;
* Contraindication to AZM use including known hypersensitivity to AZM, erythromycin, any macrolide, or ketolide drug, patients with significant hepatic impairment (direct bilirubin >1.5 mg/dL or ALT ≥ 10 times the upper limits of normal);
* Patients with known cardiac disease, cardiac arrhythmia or with electrocardiogram QT interval corrected for heart rate (QTc) ≥ 450 milisecond (ms);
* Intensive respiratory support greater than 48 hours prior to ICU admission;
* Chronic ventilation or supplemental oxygen need at home;
* Immunosuppressive conditions such as those post heart or hematopoietic stem cell transplant or receiving chemotherapy and chronic steroids;
* History of pyloric stenosis;
* AZM is deemed necessary for clinical treatment (for instance, if patient has pertussis).

Ages: 3 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 370 (Estimated)
Dates: Start 2022-02-27 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Length of Hospitalization | At discharge (Approximately 2 weeks)
  Duration of hospitalization in days for enrolled subjects

SECONDARY OUTCOMES:
Duration of oxygenation | At discharge (Approximately 1 week)
  Duration of oxygenation in days for enrolled subject
Length of ICU stay | At ICU discharge (Approximately 1 week)
  Duration of ICU stay in days for enrolled subjects

CONTACTS AND LOCATIONS:
Overall Officials: Michele Kong, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (15):
- United States (15):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Health, Indianapolis, Indiana
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma Health Sciences, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
To be determined.